CLINICAL TRIAL: NCT06494670
Title: Trends in Prevalence of 11 Site-specific Musculoskeletal Pain Among U.S. Adults, 1999-2018: a Cross-sectional Study
Brief Title: Trends in Prevalence of 11 Site-specific Musculoskeletal Pain Among U.S. Adults, 1999-2018
Status: Enrolling by invitation | Type: Observational
Sponsor: Fan luying (Other)
Responsible Party: Sponsor-Investigator, Fan luying, Investigator, Central South University
Organization: Central South University (Other)
Other Study IDs: CSU202407; 82173608 (Other Grant/Funding Number: National Natural Science Foundation of China); 81974019 (Other Grant/Funding Number: National Natural Science Foundation of China); 2022JJ40207 (Other Grant/Funding Number: Natural Science Foundation of Hunan Province of China)
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Musculoskeletal Pain; Neck Pain; Low Back Pain; Joint Pain; Shoulder Pain
Keywords: Musculoskeletal pain; Prevalence; Age-period-cohort effects
MeSH Terms: conditions — Musculoskeletal Pain; Neck Pain; Low Back Pain; Arthralgia; Shoulder Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — This study was a cross-sectional study with no intervention for participants

SUMMARY:
The goal of this observational study is to explore the prevalence trends of 11 site-specific musculoskeletal pain from 1999 to 2018. The main question it aims to answer is:

Does the prevalence of musculoskeletal pain among U.S. adults changed from 1999 to 2018? What are the trends?

Participants will answer survey questions about their musculoskeletal pain on the past three months.

DETAILED DESCRIPTION:
Musculoskeletal (MSK) pain refers to pain, either acute or chronic, affecting muscles, bones, joints, tendons, and even nerves. Common types include low back pain, neck pain, and the pain associated with osteoarthritis. These pains are the leading cause of work disability, sick leave, presenteeism, and reduced productivity. MSK pain is the leading cause of disability in the United States in 2021, ranking first in years lived with disability and fourth in disability-adjusted life years. Moreover, MSK pain is often chronic and progressive, placing a considerable strain on healthcare systems and financial resources. Estimates of US healthcare spending in 2016 revealed that low back and neck pain had the highest costs, at $134.5 billion, followed by other MSK pain, which accounted for $129.8 billion.

As the U.S. population ages, the prevalence of MSK issues may rise, leading to increased demands on the healthcare system. Although the Bone and Joint Decade 2000-2010 raised awareness about the burden of MSK conditions, significant gaps in health system improvements persist. National health policies and strategies addressing MSK health as part of noncommunicable disease care remain inadequate relative to the burden of these condition such as cardiovascular disease. Achieving the 2030 Agenda for Sustainable Development and promoting health throughout life requires a renewed and sustained focus on improving MSK health at both national and global levels. Tracking the prevalence trends of MSK pain may offer valuable insights into critical public health issues, including shifts in disease burden, healthcare access, adoption of effective therapies, and reduction in the use of inappropriate or ineffective treatments. However, previous studies have mostly focused on low back pain, and neck pain. To date, very few studies have examined trends of site-specific MSK pain prevalence using national representative sample. Prevalence and trends in other sites are also important, but no relevant studies were found. The absence of such data poses challenges in accurately estimating the burden of MSK pain.

In addition, in disease trend analysis, temporal trends generally encompass multiple dimensions. For individuals with MSK pain, prevalence risk can be divided into age, period, and birth cohort effects. Age effects reflect the influence of an individual's chronological age on MSK pain prevalence. Period effects pertain to the influence of external factors on the whole population at a particular time. These factors may include changes in medical technology, public health policies, or social and economic conditions. Cohort effects reflect the impact of common experiences and exposures unique to a particular generation or birth cohort, regardless of period or age. Understanding the contribution of age-period-cohort effects and identifying potential moderating factors for each enhances comprehension of macro-level exposures, aiding in data-driven planning.

Furthermore, Healthy People 2010 and 2020, the U.S. national public health blueprint, targeted the elimination of health disparities, including those related to MSK pain, and the attainment of health equity. To assess progress toward this objective, it is crucial to evaluate disparities in MSK pain prevalence.

In this study, utilizing a large, nationally representative sample of the US population, our objective was to explore the prevalence trends of 11 site-specific MSK pain from 1999 to 2018. We also identified cohort patterns in MSK pain prevalence, isolating age, period and cohort effects. Furthermore, we also investigated these trends across various demographic factors such as race/ethnicity, gender, age, and socioeconomic status to determine whether health disparities persist.

ELIGIBILITY:
Inclusion Criteria:

* Residents of households and noninstitutional group quarters (e.g., homeless shelters, rooming houses, and group homes);
* Persons residing temporarily in student dormitories or temporary housing are sampled within the households that they reside in permanently.

Exclusion Criteria:

* Persons with no fixed household address (e.g., homeless and/or transient persons not residing in shelters);
* Active duty military personnel and civilians living on military bases, persons in long-term care institutions (e.g., nursing homes for the elderly, hospitals for the chronically ill or physically or intellectually disabled, and wards for abused or neglected children);
* Persons in correctional facilities (e.g., prisons or jails, juvenile detention centers, and halfway houses), and U.S. nationals living in foreign countries.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The National Health Interview Survey (NHIS) is a national survey conducted by the U.S. Census Bureau on behalf of the National Center for Health Statistics (NCHS). NHIS is the principal source of information on the health of the civilian noninstitutionalized population of the United States. The target population for the NHIS is the civilian noninstitutionalized population residing within the 50 states and the District of Columbia at the time of the interview. NCHS is bound by law to protect participant data, following rigorous privacy standards that have protected every NHIS participant since the first survey in 1957. Base on NHIS data, we included adults aged 18 years and older who were interviewed in a survey wave between 1999 and 2018 in this study. From the total unweighted sample of 603,140 respondents, we excluded 37,921 due to missing data on independent variables or musculoskeletal pain, resulting in an analytic sample size of 565,219.
Sampling Method: Probability Sample
Enrollment: 565219 (Estimated)
Dates: Start 1999-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Musculoskeletal pain | 1999-2018
  Participants aged 18 years or older were asked the following questions: "During the past three months, did you have [neck pain, low back pain, or jaw/front of ear pain]?" and "During the past 30 days, did you have joint pain?". Participants who answered affirmatively to joint pain were then asked to report the site of their joint pain. The options included shoulder, elbow, hip, wrist, knee, ankle, toes, and Participants aged 18 years or older were asked the following questions: "During the past three months, did you have [neck pain, low back pain, or jaw/front of ear pain]?" and "During the past 30 days, did you have joint pain?". Participants who answered affirmatively to joint pain were then asked to report the site of their joint pain. The included shoulder, elbow, hip, wrist, knee, ankle, toes, and fingers/thumb.

IPD SHARING:
Plan to Share IPD: Yes
The data utilized in this study was sourced from the National Health Interview Survey (NHIS), with the NHIS protocol having obtained approval from the NCHS Research Ethics Review Board. Additionally, written consent was secured from all participants prior to data collection. It should be noted that all data shared have been fully anonymized and do not contain any personal identifying information about the participants.
Supporting Information: Analytic Code
Time Frame: NHIS database 1999-2018 data
Access Criteria: The data used in this study was obtained from the publicly available National Health Interview Survey (NHIS) database. The NHIS is a publicly accessible resource, and researchers can freely access and use the data for their studies.
URL: https://www.cdc.gov/nchs/nhis/about_nhis.htm